CLINICAL TRIAL: NCT02240589
Title: Memantine for Neuroprotection and Cognitive Enhancement Following Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Flora Hammond, Covalt Professor & Chair, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A70-4-0791023
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Memantine; Memory
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental): 24 weeks of memantine with accelerated titration, beginning within 48 hours of injury.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): 24 weeks of placebo matched to memantine formulation, beginning within 48 hours of injury.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Day 1 to 3: 10 mg bid memantine. Day 3 to 21: 20 mg bid memantine. Day 21 to 168: 10 mg bid memantine.
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — Day 1 to 3: 10 mg bid placebo. Day 3 to 21: 20 mg bid placebo. Day 21 to 168: 10 mg bid placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if memantine can improve cognitive and neuropsychiatric outcomes after severe traumatic brain injury.

DETAILED DESCRIPTION:
This is a pilot/feasibility study of memantine in severe traumatic brain injury (TBI) persons, employing a randomized, double-blind, placebo-controlled, design. Outcome evaluations will occur after 24 weeks of treatment (on medication) and 4 weeks after treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old of age at time of enrollment
* Severe traumatic brain injury (TBI)
* Feeding access (e.g., orogastric (OG), nasogastric (NG), or percutaneous endoscopic gastrostomy (PEG) tube) permitting delivery of memantine or placebo
* Availability of legally-authorized representative (LAR) to provide consent and participate in some study activities (e.g., monitoring for side effects, providing information about the patient)

Exclusion Criteria:

* Pre-existing history of serious neurological disorder
* Pre-existing history of serious psychiatric disorder (e.g., schizophrenia)
* Anticipated poor prognosis, based on the presence of bilaterally fixed and dilated pupils, severe hemodynamic instability, severe elevations in intracranial pressure refractory to interventions, or other factors leading to a determination of a probable non-survivable injury
* Primarily penetrating mechanism of injury (e.g., gunshot wound to the head)
* Isolated epidural hematoma with anticipated good prognosis
* Low probability of participant being compliant or being able to finish study procedures (e.g., present for outcome rating) in the judgment of the investigator
* Not English speaking (due to inability to complete outcome measure)
* Medical contraindications to memantine: Severe hepatic impairment (defined as albumin > 15gm/dL, Alk Phos > 375 U/L, ALT > 150 U/L, AST > 120 U/L or bilirubin > 3mg/dL). Moderate-to-Severe renal impairment (defined as creatinine clearance < 60)
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flora Hammond, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Facilities, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 5 | 6
Completed | 3 | 4
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (2.3) | 40.83 (6.52) | 33.82 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: California Verbal Learning Test - Second Edition (CVLT-II) - Long Delay Free Recall
Description: Neuropsychological test used to assess an individual's verbal memory abilities. The California Verbal Learning Test-Second Edition (CVLT-II) Long Delay Free Recall measures total word list items recalled after a 20-minute delay. The raw score is converted to a Z-score (Mean=0; SD=1) which was used for statistical analysis. Higher scores reflect worse performance (i.e., more recall errors) on this variable.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
z-score | -2.000 (1.000) | -1.375 (2.016)

2. Secondary Outcome: CVLT-II Trials 1-5 Free Recall Total
Description: Neuropsychological test used to assess an individual's verbal memory abilities. California Verbal Learning Test-Second Edition (CVLT-II) Trials 1-5 Free Recall Total measures the sum of all word list items correctly recalled on learning trials 1 through 5. This raw score is converted to a T-score (Mean=50; SD=10) which was used for statistical analysis. The total A1-5T score reflects accurate recall over the five learning trials of the first list, and is most often used as a summary index of learning on the CVLT-II, with higher scores reflecting better performance.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
t-score | 31.000 (10.817) | 37.250 (15.262)

3. Secondary Outcome: Brief Visuospatial Memory Test - Revised (BVMT-R) Delayed Recall
Description: Brief Visuospatial Memory Test-Revised (BVMT-R) Delayed Recall measures the correctly recalled designs (i.e., standard scoring of accuracy and location as described in the manual) after a 25 minute delay. The delayed recall raw score ranges from 0 to 12 with 12 being the highest and best possible score. The raw score is converted to a T-score (Mean=50; SD=10) which was used for statistical analysis.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
t-score | 47.00 (4.583) | 45.50 (11.561)

4. Secondary Outcome: BVMT-R Learning
Description: Brief Visuospatial Memory Test-Revised (BVMT-R) Learning measures the correctly recalled designs (i.e., standard scoring of accuracy and location as described in the manual) over 3 learning trials. The Learning raw score is the sum of the higher number of correctly recalled designs on either Trial 2 or Trial 3 minus the number of correctly recalled designs on Trial 1. A higher score is a better score. The raw score was converted to a T-score (Mean=50; SD=10) for analysis.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
t-score | 60.00 (8.266) | 46.50 (1.000)

5. Secondary Outcome: Trail Making Part B
Description: Neuropsychological test of visual attention and executive functioning. The trail making tests are thought to reflect a variety of cognitive processes including attention, visual search and scanning, sequencing and shifting, psychomotor speed, abstraction, flexibility, ability to execute and modify a plan of action, and ability to maintain two trains of thought simultaneously. In Trails B, the participant is instructed to draw lines to connect numbers and letters in an alternating numeric and alphabetic sequence as rapidly as possible. Lower scores are better scores and the range of scores can be from 0 to no limit for Trail Making Test part B. This is a timed test and the number of seconds to complete the task is recorded. The unit of measure in seconds is converted to a scaled score (mean =10, SD = 3) using the Heaton et al. norms with lower scores indicating better performance.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: scaled score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
scaled score | 11.67 (6.351) | 13.25 (4.349)

6. Secondary Outcome: Stroop Interference
Description: Stroop Interference Test is a neuropsychological test to assess a person's executive function. Specifically, the test is thought to reflect selective attention, cognitive flexibility and processing speed. The raw score for this measure is the number of items correctly identified within 45 seconds. The raw score was converted to a T-score (mean=50; SD=10) for analysis. Higher scores reflect better performance and less interference on reading ability.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
t-score | 51.67 (6.807) | 52.25 (7.320)

7. Secondary Outcome: Behavior Rating Inventory of Executive Function (BRIEF) Inhibit
Description: The Behavior Rating Inventory of Executive Function (BRIEF) Inhibit subscale is a rating scale completed by the participant and independently by an observer that assesses the ability to control impulses (inhibitory control) and to stop engaging in a behavior. The frequency of behaviors indicated by items is rated on a 3-point scale (never, sometimes, often). The raw score for the Inhibit subscale is the sum of ratings for the 8 items included in this measure. This sum was converted to a T-score (mean=50; SD=10) for analysis. Higher scores suggest a higher level of dysfunction in a specific domain of executive functions.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
t-score | 46.00 (9.416) | 61.00 (17.569)

8. Secondary Outcome: Traumatic Brain Injury Quality of Life Anger (TBI QOL Anger)
Description: The TBI-QOL Anger item bank includes 38 hierarchically ordered items designed to measure the full continuum of anger in a way which is both sensitive and appropriate for TBI. The TBI-QOL Anger item bank can be administered as a computer-adaptive test (CAT), allowing precise measurement of self-reported anger using only 4-8 adaptively selected items. Using CAT technology, an individual participant's responses to the TBIQoL Anger scale generated a T-score (Mean=50; SD=10) with a range of 0 (lowest anger) to 100 (greatest anger).
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: scaled score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 3 | 4
scaled score | 49.725 (8.684) | 45.375 (9.854)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Memantine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=5) | Placebo (N=6)
Death due to withdrawal of care (Nervous system disorders) | 0 (0) | 1 (1) — withdrawal of care
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=5) | Placebo (N=6)
Intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Conjuectivitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Other, infection (Infections and infestations) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
emesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neurostorming (Nervous system disorders) | 3 (3) | 2 (2)
Agitation (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
seizures (Nervous system disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
lethargy (Nervous system disorders) | 0 (0) | 1 (1)
fatigue (Nervous system disorders) | 1 (1) | 0 (0)
insomnia (Nervous system disorders) | 1 (1) | 2 (2)
dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
pain (Nervous system disorders) | 2 (2) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypophosphotemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No